CLINICAL TRIAL: NCT02714634
Title: Randomized Controlled Clinical Trial Evaluating Methotrexate or Leflunomide + Targeted Therapy Versus Methotrexate or Leflunomide + Sulfasalazine + Hydroxychloroquine in Patients With Rheumatoid Arthritis and Insufficient Response to Methotrexate or Leflunomide
Brief Title: Clinical Trial Evaluating Methotrexate or Leflunomide + Targeted Therapy Versus Methotrexate or Leflunomide + Sulfasalazine + Hydroxychloroquine in Patients With Rheumatoid Arthritis and Insufficient Response to Methotrexate or Leflunomide
Acronym: BIO3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6020
Record Dates: First submitted 2016-02-01; First posted 2016-03-21 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis; Insufficient Response to Methotrexate or Leflunomide
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Leflunomide; Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- methotrexate + targeted therapy group (Experimental): Methotrexate or leflunomide +
  targeted therapy chosen by investigator
  Interventions: Drug: Methotrexate + targeted therapy administration
- Triple therapy (Active Comparator): Triple therapy using 3 conventional disease modifying drugs (DMARDs)
  Interventions: Drug: methotrexate or leflunomide + sulfasalazine + hydroxychloroquine administration

INTERVENTIONS:
Drug: Methotrexate + targeted therapy administration — * Methotrexate or leflunomide + adalimumab or
  * Methotrexate or leflunomide + certolizumab or
  * Methotrexate or leflunomide + etanercept or
  * Methotrexate or leflunomide + golimumab or
  * Methotrexate or leflunomide + infliximab or
  * Methotrexate or leflunomide + abatacept or
  * Methotrexate or leflunomide + rituximab or
  * Methotrexate or leflunomide + tocilizumab or
  * Methotrexate or leflunomide + sarilumab or
  * Methotrexate or leflunomide + filgotinib or
  * Methotrexate or leflunomide + upadacitinib or
  * Methotrexate or leflunomide + Tofacitinib or
  * Methotrexate or leflunomide + baricitinib
  Arms: methotrexate + targeted therapy group
Drug: methotrexate or leflunomide + sulfasalazine + hydroxychloroquine administration
  Arms: Triple therapy

SUMMARY:
Approximately, 40 to 50% of patients with rheumatoid arthritis (RA), the most frequent inflammatory arthritide, are non responders to the consensual 1st line of treatment : methotrexate. In these patients, it is well demonstrated that the addition of other immunomodulatory drug(s) often results in a significant improvement. However, the best option regarding the drug(s) to add remains unclear. Rheumatologists are currently used to adding a targeted therapy, such as anti-TNFα, and more recently abatacept or tocilizumab. Triple therapy using 3 conventional disease-modifying drugs (DMARDs), methotrexate or leflunomide+salazopyrine+hydroxychloroquine could be an alternative option to targeted therapies, all the more as they have a more favorable safety profile and a much lower cost. Uncertainty remains regarding the superiority of targeted therapies on triple therapy in methotrexate or leflunomide insufficient responders (IR). Investigators decided to address this issue by performing a randomized controlled pragmatic trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient with rheumatoid arthritis according to EULAR/ACR 2010 criteria
* DAS28-CRP>3.2
* Insufficient response to methotrexate at a weekly dose≥15mg after at least 3 months or to leflunomide at a dose of 10 (in case 20 mg are not well tolerated) to 20 mg per day after 3 months of treatment
* RA radiographic erosions and/or serum rheumatoid factor associated to anti-Cyclic Citrullinated Peptide (Anti-CCP)
* Age greater or equal to 18 years
* Written informed consent, dated and signed before initiating any trial-related procedure
* Affiliation to a social insurance system
* Women of child bearing potential, negative β-HCG assay (Human chorionic gonadotropin)
* Effective method of birth control during the study and continuing after the discontinuation of the investigational drug or study. The duration will depend on the drug used (referred to the summary product characteristic).

Exclusion Criteria:

* Previous treatment with or contraindication to targeted therapies (biologic or JAK/STAT inhibitor)
* Previous treatment with triple therapy
* Other inflammatory arthritis except RA associated with Sjögren's syndrome
* Contraindication to all biologics/ JAK/STAT inhibitors or to methotrexate, leflunomide, sulfasalazine and hydroxychloroquine
* Corticosteroids at a dose >15 mg/d of equivalent prednisone for at least 4 weeks before the inclusion
* Absence of tuberculosis screening
* Patient who cannot be followed during 12 months
* Pregnancy, breastfeeding, desire of pregnancy in the 12 months
* Drug addiction, addiction to alcohol
* Participation in a clinical study with an investigational product within 4 weeks prior to the start of the study treatment
* Women of child bearing potential, unless they are using an effective method of birth control
* Patient under law protection
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2016-03-30 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Numbers of participant with low disease activity (DAS28-CRP<3.2) and a daily dose ≤ 7.5 mg/day of equivalent prednisone | At 12 months

SECONDARY OUTCOMES:
Serious adverse events rate | At 3, 6, 9 and at 12 months
Blood concentrations of hydroxychloroquine, leflunomide, sulfasalazine and methotrexate in the triple therapy group and methotrexate, leflunomide, biologic / JAK/STAT inhibitor and anti-drug antibody in the other group. | at 6, and 12 months
Clinical disease activity index (CDAI). | At inclusion, 3, 6, 9 and 12 months
DAS 28 CRP score. | at inclusion, 3, 6, 9 and 12 months.
2010 ACR (American College of Rheumatology)/EULAR classification Criteria for RA, ACR 20, 50, 70 and boolean remission. | at 3, 6, 9 and 12 months.
Modified Sharp Van der Heijde score. | at inclusion and at 12 months
Change in comedications (dose) | at 3, 6, 9 and 12 months
Change in comedications (route of administration) | at 3, 6, 9 and 12 months
Change in comedications (drug) | at 3, 6, 9 and 12 months
QUALISEX score at inclusion, 6 months and at 12 months. | at inclusion, 6 months and at 12 months.
Medico-economic costs. | at inclusion, 3, 6, 9 and at 12 months.
Treatment compliance | at 3, 6, 9 and 12 months
  A questionnaire will be filled by patient

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No